CLINICAL TRIAL: NCT05603676
Title: Intermittent Hypoxia-hyperoxia Conditioning as a New Therapeutic Intervention to Reduce Hypertension
Brief Title: Intermittent Hypoxia-hyperoxia Conditioning as a New Therapeutic Intervention to Reduce Hypertension (HyperIHHC)
Acronym: HyperIHHC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Gregoire Millet (Other)
Collaborators: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Sponsor-Investigator, Gregoire Millet, Associate professor, University of Lausanne
Organization: University of Lausanne (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-01295
Record Dates: First submitted 2022-09-20; First posted 2022-11-03 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-10

CONDITIONS: Hypertension
Keywords: Intermittent hypoxia-hyperoxia conditioning; Vascular function; Hemorheology
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: This project is a single center national study. It is designed as a randomized single-blinded parallel group control study. Single-blinded means that participants will not be inform than a half will follow a placebo intervention. Parallel group means that the design serves to compare different experimental conditions. Randomized means that the participants are assigned to the two different conditions randomly (by chance alone). Control means that one of the group/conditions is the standard of comparison (control participant achieving placebo and IHHC interventions). A follow-up, one month after the intervention will be done.
Who Masked: Participant
Masking Description: Single-blinded means that participants will not be inform than a half will follow a placebo intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Hypertensive IHHC (Experimental): Hypertensive participants who performed IHHC
  Interventions: Other: Intermittent hypoxia-hyperoxia conditioning
- Hypertensive placebo (Placebo Comparator): Hypertensive participants who performed placebo intervention
  Interventions: Other: Placebo intervention
- Healthy IHHC (Active Comparator): Healthy participants who performed IHHC
  Interventions: Other: Intermittent hypoxia-hyperoxia conditioning
- Healthy Placebo (Sham Comparator): Healthy participants who performed placebo intervention
  Interventions: Other: Placebo intervention

INTERVENTIONS:
Other: Intermittent hypoxia-hyperoxia conditioning — The IHHC protocol consist of 6 bouts of 6 min breathing hypoxia (FiO2 = 11.5%) following by 3 min breathing hyperoxia (FiO2 = 31.5%) (Figure 2). The total duration of a session is 54 minutes. Participant will undergo 3 session a week for 6 weeks. During the session, participant will be comfortably seated on an armchair and equipped with a mask and a non-rebreathing valve rely to a motorized valve that blindly change the gas input from two different mixing chambers with hypo and hyperoxic gas mixture. Participants will be instructed to relax and breath normally throughout the session.
  Arms: Healthy IHHC; Hypertensive IHHC
Other: Placebo intervention — Placebo intervention will be like the IHHC protocol but with mixing chambers full of ambient air. The total duration of a placebo session is 54 minutes. Participant will undergo 3 session a week for 6 weeks. During the session, participant will be comfortably seated on an armchair and equipped with a mask and a non-rebreathing valve rely to a motorized valve that blindly change the gas input from two different mixing chambers with ambient air. Participants will be instructed to relax and breath normally throughout the session.
  Arms: Healthy Placebo; Hypertensive placebo

SUMMARY:
The primary objective of this project is to examine the efficiency of intermittent hypoxia-hyperoxia conditioning (IHHC) protocol to improve vascular health and reduce blood pressure in hypertensive patients (stage 1). The result of the present study will investigate if IHHC could be a therapeutic treatment for hypertensive individuals. The investigation is designed with a placebo intervention (air ambient) and a control group (age-matched healthy participants). The interest of short cycles of intermittent hypoxia-hyperoxia is due to the triggering of the vasodilatory response in a greater extent compared to the pressor mechanisms since the exposure duration remains short. Therefore, it can be hypothesized that control and hypertensive groups achieving IHHC may exhibit a decreased blood pressure compared to the control and hypertensive groups achieving placebo intervention. The control group may show greater change than hypertensive due to higher vascular reserve.

The secondary objective of the study is to understand the underlying mechanism of the beneficial effects of IHHC, especially the role of blood hemorheological changes. Based on available literature, it is know that hypoxia induce an increase in blood viscosity. One may hypothesize that with such a short hypoxic dose used during IHHC, only minor change in blood viscosity may occur. However, a slight rise in blood viscosity is known to stimulate NO synthase and then to produce more NO. Hence it could be one of the mechanisms involved in the early vasodilatory response to hypoxia. These findings are in line with the reported higher NO end-product metabolites during exercise in normoxia and hypoxia in subjects who showed a rise in blood viscosity after exercise. The hypothesis is that the magnitude of IHHC beneficial effects is related to change in blood viscosity and its determinants.

DETAILED DESCRIPTION:
The prevalence and absolute burden of hypertension is rising worldwide and represents one of the leading modifiable risk factors for cardiovascular diseases being indirectly involved in the development of, for instance, stroke, kidney diseases, and dementia.

There is rather solid evidence supporting the assumption that intermittent and continuous hypoxia at rest or in combination with exercise is generally effective to reduce blood pressure and positively influence vascular health.

A well-designed and controlled hypoxic stimulus may induce benefits for health and is known as hypoxia conditioning (HC). Indeed, brief and repeated exposures to hypoxia trigger cellular and systemic physiological adaptations that make the organism more resilient to subsequent severe hypoxic stress, and possibly also to other stressors.

The mechanisms associated with an antihypertensive effect of moderate hypoxia may include vascular adaptions (e.g. increased vascularisation and endothelium-dependent vasodilatation) as well as adaptations in the autonomic nervous system (e.g. reduced sympathetic activity).

Hypoxia exposure leads to a multiphasic blood flow and pressure response over time. The first and immediate phase following hypoxic stimulus is characterized by a systemic vasodilation that aims to counteract the decrease in arterial oxygen (O2) content and subsequent peripheral O2 delivery. If hypoxia exposure lasts for more than few minutes, pressor mechanisms, such as sympathetic activation, a rise in arterial stiffness, an increase in endothelin-1 levels, a baroreflex dysfunction and an elevation in blood viscosity, exceed vasodilatory responses resulting in a rise of blood pressure. However, the mechanisms at the onset of the early blood pressure response are beneficial for vascular health and an improvement in vascular function following intermittent hypoxia exposure has been reported during both intermittent resting exposure (FiO2: 10-14%, 3-5 minutes of normobaric hypoxia per cycle, 3-25 cycles/day during 10 to 30 days [7]) or intermittent exposure combined with exercise (2 hrs of hypobaric hypoxic exposure (FiO2: 16.5%) with 30 minutes of moderate intensity exercise, 4 days/week during 8 weeks).

This is likely related to the release of vasodilatory molecules, mainly nitric oxide (NO), and the activation of transcriptional factors, such as hypoxia inducible factor (HIF-1) and nuclear factor erythroid-2 related factor 2 (Nrf2), which are beneficial for vascular function through the enhanced production/activity of vascular endothelial growth factor, erythropoietin, and antioxidant enzymes. However, it was reported that severe hypoxia (FiO2 = 12%) but not moderate hypoxia (FiO2 = 15%) (1 h/day, 5 days/week for 4 weeks) impaired endothelial function [19] suggesting that vascular benefits from hypoxia are a matter of dose.

Cardiovascular disorders are associated with poor vascular function, increased arterial stiffness or impaired endothelial and non-endothelial flow-mediated dilation. Although less investigated, blood flow properties also play a key role in the development and progression of vascular disorders and dysfunction. More particularly, the viscosity of blood has a major impact on regulating vascular function. One of the most famous hematological adaptations following chronic hypoxia exposure is the increase in total hemoglobin mass, generally associated to the elevation in hematocrit (Hct), which may enhance the oxygen-carrying capacity. However, Hct is also a major determinant of blood viscosity, and any elevation in blood viscosity may have consequences on vascular resistance and blood perfusion, particularly in the absence of compensatory mechanisms. Hence, in order to understand the benefits of hypoxia exposure on vascular health, the related changes in blood viscosity must be considered. Unfortunately, studies on hypoxia conditioning and vascular functions usually do not measure the change in blood viscosity, which remains a forgotten factor for the understanding of hypoxia-related improvement/impairment of vascular function.

An innovative strategy of conditioning is to interspersed hypoxia exposure trial with hyperoxic one, since the latter also stimulate HIF-1 and Nfr2 pathway, and is called intermittent hypoxia/hyperoxia conditioning (IHHC). Three studies have found that IHHC can decrease systolic (- 2.9% to - 13.9%) and diastolic blood pressure (- 9.0% to 14.0%), although the changes did not always reach statistical significance (p=0.07). With regard to studies using intermittent hypoxia/normoxia, young males with stage I hypertension were exposed to 20 consecutive days of intermittent hypoxic exposure (4-10 cycles per session, 3 min of hypoxia [ FiO2 = 10%] interspersed by 3 min of normoxia). A decrease of 22 mmHg in systolic and 16.6 mmHg in diastolic blood pressure was reported after exposure. A decreases of 10-30 mmHg in systolic and 10-15 mmHg in diastolic blood pressure in patients with stage I to II hypertension after intermittent or prolonged hypoxic exposure was also reported. Recent meta-analysis have shown that every reduction of 10 mmHg in systolic or 5 mmHg in diastolic blood pressure reduced the risk of major cardiovascular events by 20%, the genesis of cardiovascular diseases by 17-40%, and all-cause mortality by 13%. Indeed, a decrease of even 2 mmHg in systolic blood pressure would involve a 10% lower stroke mortality and about 7% lower mortality for cardiovascular heart diseases or other vascular causes in middle age. Given the evidence that IHHC can trigger a reduction in systolic and diastolic blood pressure in patients with and without cardiovascular diseases, it can be considered as a promising therapeutic strategy to reduce systemic blood pressure. Therefore, the hypotensive effect of IHHC is practically relevant to prevent the genesis or exacerbation of cardiovascular diseases and ensure a healthy life.

The primary objective of this project is to examine the efficiency of IHHC protocol to improve vascular health and reduce blood pressure in hypertensive patients (stage 1). The result of the present study will investigate if IHHC could be a therapeutic treatment for hypertensive individuals. The investigation is designed with a placebo intervention (air ambient) and a control group (age-matched healthy participants). The interest of short cycles of intermittent hypoxia-hyperoxia is due to the triggering of the vasodilatory response in a greater extent compared to the pressor mechanisms since the exposure duration remains short. Therefore, it can be hypothesized that control and hypertensive groups achieving IHHC may exhibit a decreased blood pressure compared to the control and hypertensive groups achieving placebo intervention. The control group may show greater change than hypertensive due to higher vascular reserve.

The secondary objective of the study is to understand the underlying mechanism of the beneficial effects of IHHC, especially the role of blood hemorheological changes. Based on available literature, it is know that hypoxia induce an increase in blood viscosity. One may hypothesize that with such a short hypoxic dose used during IHHC, only minor change in blood viscosity may occur. However, a slight rise in blood viscosity is known to stimulate NO synthase and then to produce more NO. Hence it could be one of the mechanisms involved in the early vasodilatory response to hypoxia. These findings are in line with the reported higher NO end-product metabolites during exercise in normoxia and hypoxia in subjects who showed a rise in blood viscosity after exercise. The hypothesis is that the magnitude of IHHC beneficial effects is related to change in blood viscosity and its determinants.

ELIGIBILITY:
Inclusion Criteria:

1. to be aged between 44 and 65 years old.
2. for women, post-menopausal will be considered.
3. for hypertensive group, stage 1 hypertension: systolic blood pressure (140-159 mmHg) and/or diastolic blood pressure (90-99 mmHg).
4. free of other disease than hypertension and free of anti-hypertensive treatment medication.
5. Hypertensive participants with 14 days of hypertensive drugs wash-out.
6. able to complete all sessions.
7. able to give consent.

Exclusion Criteria:

1. Peripheral arterial disease
2. Atrial fibrillation
3. Hypoxic congenital heart diseases
4. Pulmonary Hypertension
5. using dietary supplements or drugs which interfere with the measurements (nitrate supplementation)

Ages: 44 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2022-11-15 (Estimated); Primary Completion 2023-05-15 (Estimated); Study Completion 2023-05-15 (Estimated)

PRIMARY OUTCOMES:
24 hours Blood pressure change form pre to post intervention | One week before the intervention and one week after the intervention
  a major risk factor, when too high, for cardiovascular diseases will be continously measured for 24 hours.

SECONDARY OUTCOMES:
Baroreflex sensitivity | One week before the intervention and one week after the intervention
  a measurement of the mechanism that regulates acute blood pressure changes via controlling heart rate, contractility, and peripheral resistance. It is based on the quantification of RR interval changes related to blood pressure changes [ms/mmHg]. Alterations of the BRS contribute to the development and progression of cardiovascular diseases.
Reactive hyperemia index | One week before the intervention and one week after the intervention
  a measure for arterial endothelial function
Vascular occlusion test (VOT) | One week before the intervention and one week after the intervention
  an investigation of microvascular function. The combination of near infrared spectroscopy (NIRS) with the VOT has emerged as a noninvasive tool for the evaluation of downstream microvascular responses to ischemia/reperfusion through the NIRS-VOT-derived reperfusion slope
Pulse wave velocity | One week before the intervention and one week after the intervention
  calculated by the delay between two pulse waves, this index reflects arterial stiffness.
Cerebrovascular reactivity to carbon dioxide (CO2) | One week before the intervention and one week after the intervention
  a measurement of the mechanism regulating cerebral blood flow. It is based on the change in carotid artery velocity when cerebral vasoactive substance (CO2) is manipulated, i.e., hypercapnia and hypocapnia.
Advanced oxidation protein products | One week before the intervention and one week after the intervention
  Marker of protein oxidation
Malondialdehyde | One week before the intervention and one week after the intervention
  Markers of lipid oxidation
Superoxide dismutase | One week before the intervention and one week after the intervention
  An antioxydant enzyme
Glutathion peroxydase | One week before the intervention and one week after the intervention
  An antioxydant enzyme
Catalase | One week before the intervention and one week after the intervention
  An antioxydant enzyme
Nitric oxide end products | One week before the intervention and one week after the intervention
  A marker of NO metabolism and oxidation
Blood viscosity (cp) | One week before the intervention and one week after the intervention
  Blood viscosity at native hematocrit will be measured at high and low shear rate
Blood volume | One week before the intervention and one week after the intervention
  a measure of the total amount of blood volume which is necessary to better understand the vascular and hemorheological changes
Plasma viscosity (cp) | One week before the intervention and one week after the intervention
  Plasma viscosity will be measured at high shear rate
Hematocrit | One week before the intervention and one week after the intervention
  will be measured by flow cytometry

CONTACTS AND LOCATIONS:
Overall Officials: Grégoire P Millet, PhD, Principal Investigator — University of Lausanne
Locations (1):
- ISSUL, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lyamina NP, Lyamina SV, Senchiknin VN, Mallet RT, Downey HF, Manukhina EB. Normobaric hypoxia conditioning reduces blood pressure and normalizes nitric oxide synthesis in patients with arterial hypertension. J Hypertens. 2011 Nov;29(11):2265-72. doi: 10.1097/HJH.0b013e32834b5846. PMID 21897291
- [Background] Ettehad D, Emdin CA, Kiran A, Anderson SG, Callender T, Emberson J, Chalmers J, Rodgers A, Rahimi K. Blood pressure lowering for prevention of cardiovascular disease and death: a systematic review and meta-analysis. Lancet. 2016 Mar 5;387(10022):957-967. doi: 10.1016/S0140-6736(15)01225-8. Epub 2015 Dec 24. PMID 26724178
- [Background] Serebrovskaya TV, Xi L. Intermittent hypoxia training as non-pharmacologic therapy for cardiovascular diseases: Practical analysis on methods and equipment. Exp Biol Med (Maywood). 2016 Sep;241(15):1708-23. doi: 10.1177/1535370216657614. Epub 2016 Jul 12. PMID 27407098